CLINICAL TRIAL: NCT05268510
Title: Phase IIA Trial of Short-term Chemotherapy and Pembrolizumab, Followed by Pembrolizumab and Olaparib As Firstline Therapy in Her-2 Negative Gastric/gastroesophageal-junction (GEJ) Adenocarcinoma
Brief Title: Chemotherapy and Pembrolizumab, Followed by Pembrolizumab and Olaparib As Firstline Therapy in Her-2 Negative Gastric/GEJ Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLESTAR
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Esophagogastric Adenocarcinoma
Keywords: gastric adenocarcinoma; GEJ adenocarcinoma; Her-2 negative esophagogastric adenocarcinoma
MeSH Terms: interventions — pembrolizumab; olaparib

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive 2 six-week (q42d) cycles of mod. FOLFOX-6 plus 400 mg pembrolizumab. Alternatively, subjects may receive 2 six-week (q42d) cycles of CAPOX plus 400 mg pembrolizumab. The decision for either mod. FOLFOX-6 or CAPOX is made at the sole discretion of the investigator taking into account the best interest of the patient.
  Following the chemotherapy induction phase, the subjects are scheduled to receive up to 16 six-week (q42d) cycles of pembrolizumab (400 mg) plus olaparib (300 mg bid.).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy plus Pembrolizumab followed by Pembrolizumab and Olaparib (Experimental): Chemotherapy plus Pembrolizumab 2 cycles à 6 weeks:
  Pembrolizumab+mod FOLFOX-6:
  * Pembrolizumab 400 mg 30 min. day 1
  * Oxaliplatin 85 mg/m² 2h day 1, 15, 29
  * Leucovorin 400 mg/m² 2h day 1, 15, 29
  * 5-FU 400 mg/m² bolus, followed by 2.400 mg/m² 46h day 1, 15, 29
  or
  Pembrolizumab+CapOx:
  * Pembrolizumab 400 mg 30 min. day 1
  * Oxaliplatin 130 mg/m² 2h day 1,22
  * Capecitabine 1.000 mg/m² bid. day 1-14, 22-35
  Consolidation phase Pembrolizumab and Olaparib max 16 cycles à 6 weeks:
  * Pembrolizumab 400 mg 30 min. day 1
  * Olaparib 300 mg bid. cont. day 1 to 42
  Interventions: Drug: Pembrolizumab; Drug: Olaparib; Drug: mFOLFOX-6; Drug: CapOX

INTERVENTIONS:
Drug: Pembrolizumab — 400 mg Pembrolizumab day 1 Q6W (max. 18 cycles)
  Other Names: Keytruda
Drug: Olaparib — 300 mg Olaparib bid. cont. day 1 to 42 (max. 16 cycles)
  Other Names: Lynparza
Drug: mFOLFOX-6 — Oxaliplatin 85 mg/m² 2h day 1, 15, 29 plus Leucovorin 400 mg/m² 2h day 1, 15, 29 plus 5-FU 400 mg/m² bolus, followed by 2.400 mg/m² 46h day 1, 15, 29; Q6W, 2 cycles
Drug: CapOX — Oxaliplatin 130 mg/m² 2h day 1,22 plus Capecitabine 1.000 mg/m² bid. day 1-14, 22-35; Q6W, 2 cycles

SUMMARY:
This is a multicenter, single arm, prospective, open-label phase II trial investigating the clinical activity of a first-line therapy consisting of induction chemotherapy plus pembrolizumab (12 weeks of mod. FOLFOX-6 plus pembrolizumab or 12 weeks of CAPOX plus pembrolizumab) followed by pembrolizumab plus olaparib.

DETAILED DESCRIPTION:
Her-2 negative patients suffering from metastatic or unresectable gastric/GEJ adenocarcinoma will be included in the study. Eligible subjects will receive 2 six-week (q42d) cycles of mod. FOLFOX-6 plus pembrolizumab. Alternatively, subjects may receive 2 six-week (q42d) cycles of CAPOX plus pembrolizumab. The decision for either mod. FOLFOX-6 or CAPOX is made at the sole discretion of the investigator taking into account the best interest of the patient. Following the chemotherapy induction phase, the subjects are scheduled to receive pembrolizumab plus olaparib until tumor progression or occurrence of limiting toxicity for a maximum of 16 cycles (q42d, total 18 cycles, approx. 2 years).

The primary objective of this phase II study is to assess the overall survival at 1 year. Secondary objectives are the assessment of the objective response rate, the best overall response, progression-free survival, overall survival and treatment feasibility rate along with safety and toxicity of the treatment.

The exploratory objective is to assess whether clinical efficacy correlates with molecularly-defined subgroups (PD-L1 expression, HR alterations, MSI subtypes, and others).

The study will be accompanied by an explorative translational research analysis of blood and tumor samples.

The compositional changes of leukocyte states and their gene expression changes under combination immunotherapy will be analyzed using single cell RNA sequencing. Using factor analysis methods, we will analyze the environmental cues shaping leukocyte states and compare these features in responders and non-responders to therapy and correlate these with overall and progression-free survival. In addition, centralized PD-L1 expression and molecular sequencing of tumor tissue will be performed with a focus on alterations of HRD pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or unresectable, histologically confirmed Her-2 negative (as assessed locally by a certified test) adenocarcinoma of the gastroesophageal junction (AEG I- III according to Sievert´s classification) or the stomach.
2. Adjuvant/neoadjuvant or perioperative chemotherapy or chemoradiotherapy must have been finished at least 6 months before start of the study intervention.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Ability for oral intake of the study drug.
5. Male/female* participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of esophagogastric adenocarcinoma will be enrolled in this study.

   * There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.
6. Male participants: A male participant must agree to use a contraception during the treatment period and for at least 6 months after the last dose of study intervention and refrain from donating sperm during this period.
7. Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 6 months after the last dose of study intervention.
8. The participant provides written informed consent for the trial.
9. Have measurable or evaluable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
10. Have provided archival tumor tissue sample. FFPE tissue blocks are preferred to slides.
11. Have adequate organ function as defined in the following table. Specimens must be collected within 14 days prior to the start of study intervention:

Hematological:

* Absolute neutrophil count (ANC) ≥ 1500/µL
* Platelets ≥ 100 000/µL
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L(a)

Renal:

* Measured or calculated (b) creatinine clearance≥ 50 mL/min

Hepatic:

* Total bilirubin ≤ 1.5 ×ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases)

Coagulation

* International normalized ratio (INR) OR prothrombin time (PT)
* Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within the last 2 weeks.
2. Creatinine clearance (CrCl) should be calculated per institutional standard.

   Exclusion Criteria:
   1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to start of study intervention. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
   2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137). Has received any previous treatment with a PARP inhibitor, including Olaparib.
   3. Has received prior systemic anti-cancer therapy for metastatic or locally advanced (irresectable) disease. A prior neoadjuvant or adjuvant chemotherapy is allowed (see inclusion criterion 2)
   4. Persistent clinically relevant toxicities, CTCAE Grade > 2 caused by previous cancer treatment.
   5. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
   6. Participant received colony-stimulating factors (eg, granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM CSF] or recombinant erythropoietin) within 28 days prior to the first dose of study intervention.
   7. Participant is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption.
   8. Major surgery within 2 weeks of starting study intervention and patients must have recovered from any effects of any major surgery.
   9. Participant is currently receiving either strong (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil) inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study. The required washout period prior to starting olaparib is 2 weeks. Note: a current list of strong/moderate inhibitors of CYP3A4 can be found at the following website: https://www.fda.gov/drugs/drug-interactions-labeling/drug- development-and-drug-interactions-table-substrates-inhibitors-and-inducers
   10. Participant is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (eg. bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study. The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.

       Note: a current list of strong/moderate inducers of CYP3A4 can be found at the following website: https://www.fda.gov/drugs/drug-interactions-labeling/drug- development-and-drug-interactions-table-substrates-inhibitors-and-inducers
   11. Concomitant use of drugs inhibiting DPD activity (including sorivudine, brivudine), the required wash out phase is 4 weeks before start of the study intervention.
   12. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
   13. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
   14. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
   15. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
   16. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
   17. Participant has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
   18. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously completely resected brain metastases may participate if there is no sign of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
   19. Has severe hypersensitivity (≥ Grade 3) to FOLFOX or CAPOX-based chemotherapy, olaparib, pembrolizumab and/or any of its excipients.
   20. Known DPD deficiency. Patients with a reduced DPD activity (CPIC activity score of 1.0-1.5) might participate in the study and receive a reduced dosage of 5- FU/capecitabine after discussion with the coordinating investigator and sponsor [https://cpicpgx.org/guidelines/guideline-for-fluoropyrimidines-and-dpyd/]
   21. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
   22. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
   23. Has an active infection requiring systemic therapy.
   24. Has a known history of Human Immunodeficiency Virus (HIV) infection (known HIV1/HIV2 antibodies positive).
   25. Has a known history of/active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
   26. Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan, previous allogenic bone marrow/blood transplantation or any psychiatric disorder or substance abuse that prohibits obtaining informed consent.
   27. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 6 months after the last dose of study intervention.
   28. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) rate at 1 year | 1 year after enrolment
  Overall survival (OS) rate at 1 year defined as the percentage of patients who remain alive one year after enrollment into the study

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 55 months
  Progression-free survival (PFS), defined as time from enrollment to disease progression according to RECIST 1.1 and iRECIST or death due to any cause
Objective response rate (ORR) | up to 55 months
  ORR - percentage of patients with complete response (CR) or partial response (PR) according to RECIST 1.1 and iRECIST.
Best Overall Response (BOR) | up to 55 months
  BOR - best response recorded from enrollment to treatment discontinuation for any reason.
Time to tumor progression (TTP) | up to 55 months
  TTP - time from enrollment to disease progression according to RECIST 1.1 and iRECIST.
Overall Survival (OS) | up to 55 months
  OS - time from enrollment to the date of death of any cause.
Feasibility rate | 36 weeks
  Feasibility rate: severe toxicity/withdrawal rate before the fourth cycle of pembrolizumab/olaparib has been completed.
Incidence and severity of adverse events | up to 29 months (18 cycles a 6 weeks plus 110 days after last treatment)
  (Serious) Adverse Events - Recorded and graded according to NCI-CTC V5.0. Occurrence of (Serious) Adverse Events at any time during the study. Description by nature (Primary System Organ Class and Preferred Term), severity and causal relationship to drug administration

OTHER OUTCOMES:
Immune cell states (exploratory translational outcome) | up to 55 months
  Identification of immune cell states changing in abundance in responders vs non-responders under Pembrolizumab/chemotherapy. The compositional changes within cellular neighborhoods will be identified using a generalized linear model with an FDR of 0.025 and the following covariates: patient ID, timepoint (1st and 2nd sampling timepoint as per study protocol).
Predictive value of PD-L1 CPS (exploratory translational outcome) | up to 55 months
  Centralized analysis of the predictive value of PD-L1 combined prognostic score (CPS).
Other exploratory translational outcomes: | up to 55 months
  * Descriptively define the dynamics of immune cell states and their factor loadings over the entire course of therapy, including consolidation therapy with Olaparib in combination with Pembrolizumab stratified by best response status (PD/SD vs PR) and by PFS and OS under Olaparib + Pembrolizumab.
  * Correlation of efficacy of consolidation therapy with molecular alterations in the HRD pathway
  * Compare mean factor loadings per patient in responders (according to RECIST 1.1) and non-responders within each major immune subset (CD4 T cells, CD8 T cells, Natural Killer cells, dendritic cells, monocytes, naïve B cells, memory B cells) using Mann-Whitney-U tests and the Benjamini-Hochberg method. For comparison within the first immune cell subset alpha will be set to 0.0125 and will be divided by 2 for every additional subset tested to not exceed an overall false discovery rate of 0.05 for all analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH; Georg Martin Haag, PD Dr., Principal Investigator — National Center for Tumor Diseases, University Hospital Heidelberg
Locations (1):
- Universitätsklinikum Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No